CLINICAL TRIAL: NCT06989268
Title: A RANDOMISED, PLACEBO-CONTROLLED, CROSSOVER STUDY TO EVALUATE THE EFFECT OF LINACLOTIDE ON COLONIC MOTILITY ASSESSED WITH INTRALUMINAL COLONIC MANOMETRY IN HEALTHY SUBJECTS
Brief Title: Effect to Linaclotide on Colonic Motility
Status: Completed | Phase: Phase 4 | Type: Interventional
Sponsor: Universitaire Ziekenhuizen KU Leuven (Other)
Responsible Party: Sponsor
Allocation: Randomized | Model: Crossover | Masking: Triple | Purpose: Other
Other Study IDs: S56101
Record Dates: First submitted 2025-05-16; First posted 2025-05-25 (Actual); Last update posted 2025-05-25 (Actual); Status verified 2024-09

CONDITIONS: Chronic Constipation
Keywords: laxatives; constipation; linaclotide
MeSH Terms: conditions — Constipation

STUDY DESIGN:
Intervention Model Description: Open-label, randomized, reader-blinded, 2-period cross-over study
Who Masked: Participant, Investigator, Outcomes Assessor
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No | US Export: No

ARMS (2):
- Linaclotide (Active Comparator): 290 μg linaclotide once daily oral administration with 125mL of water
  Interventions: Drug: Linaclotide 290 micrograms
- Placebo (Placebo Comparator): placebo, empty capsule, once daily oral administration with 125mL of water
  Interventions: Drug: Placebo

INTERVENTIONS:
Drug: Linaclotide 290 micrograms — 290 μg linaclotide once daily oral administration with 125mL of water
  Arms: Linaclotide
Drug: Placebo — Placebo, empty capsule, once daily oral administration with 125mL of water
  Arms: Placebo

SUMMARY:
This study aim was to evaluate the effect of Linaclotide, a pharmacological treatment normally used to treat functional constipation or irritable bowel syndrome with predominant constipation, on colonic motility as assessed by high-resolution colonic manometry.

DETAILED DESCRIPTION:
Rationale: Several treatments with different modes of action are currently available for chronic constipation, including the osmotic laxative polyethylene glycol (PEG), the stimulant laxative bisacodyl, the prokinetic prucalopride and the secretagogue linaclotide. In a previous study conducted in our lab (study S54750) it has been hypothesized that only bisacodyl and prucalopride activate colonic motility. However the results have demonstrated that PEG, bisacodyl and prucalopride did not differ in their effect on colonic motility index, except for bisacodyl which induced HAPCs in a greater number of healthy subjects as compared to both prucalopride and PEG. To our knowledge, the effect of linaclotide on colonic motility has never been studied in humans.

Objectives: Primary: to evaluate the effects of linaclotide as compared to placebo on motility index and on the number of colonic high amplitude propagated contractions (HAPCs) during a 8-hour intraluminal manometry in healthy subjects. Secondary: to evaluate the association between motility parameters and sensations (abdominal gas, desire to defecate, urgency to defecate and abdominal discomfort) as well as number and consistency of bowel movements.

Investigational product, dose, and mode of administration: Regimen A: 290 μg linaclotide once daily oral administration with 125mL of water. Regimen B: placebo, empty capsule, once daily oral administration with 125mL of water.

Methodology: This is randomized, placebo controlled, 2-period cross-over study investigating the effects of placebo and linaclotide on colon motility with intraluminal manometry. On each of Treatment Period, a manometry catheter will be placed in the colon under conscious sedation and the colonic pressure will be continuously measured through 8 hours after administration of each of the investigational products (Regimen A or B).

Inclusion criteria: healthy male and non-pregnant, non-breastfeeding female participants, aged 18-65 years old at the time of consent.

Exclusion criteria: use of medications within 48 h of dose initiation; structural or metabolic diseases that affect the gastrointestinal system and functional gastrointestinal disorders; previous abdominal surgery other than appendectomy, cholecystectomy, hysterectomy, or hernia repair; known illnesses such as diabetes, cardiovascular or lung disease; use of agents that influence bowel habit, i.e. anticholinergics (not including antihistamines with anticholinergic properties), spasmolytics and prokinetics in the 7 days before the study.

ELIGIBILITY:
Inclusion Criteria:

* healthy male and non-pregnant, non-breastfeeding female participants, aged 18-65 years old at the time of consent

Exclusion Criteria:

* use of medications within 48 h of dose initiation; structural or metabolic diseases that affect the gastrointestinal system and functional gastrointestinal disorders; previous abdominal surgery other than appendectomy, cholecystectomy, hysterectomy, or hernia repair; known illnesses such as diabetes, cardiovascular or lung disease; use of agents that influence bowel habit, i.e. anticholinergics (not including antihistamines with anticholinergic properties), spasmolytics and prokinetics in the 7 days before the study

Ages: 18 Years to 65 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Adult, Older Adult
Enrollment: 10 (Actual)
Dates: Start 2014-02-10 (Actual); Primary Completion 2015-02-15 (Actual); Study Completion 2015-06-03 (Actual)

PRIMARY OUTCOMES:
Colonic motor patterns during Linaclotide or Placebo administration in healthy subjects. | during a 12-hour intraluminal manometry]
  Number of colonic high amplitude propagated contractions (HAPCs)

SECONDARY OUTCOMES:
Association between motility parameters and number and consistency of bowel movements in healthy subjects | during a 12-hour intraluminal manometry]
  Number of colonic motor patterns and number of bowel movements and stool consistency assessed by Bristol Stool Chart

CONTACTS AND LOCATIONS:
Overall Officials: Jan Tack, MD PhD, Principal Investigator — Universitaire Ziekenhuizen KU Leuven

IPD SHARING:
Plan to Share IPD: No